CLINICAL TRIAL: NCT01000376
Title: An Open-Label, Phase I Study to Evaluate the Pharmacokinetics and Tolerance of Co-administration of Oral Multiple Dose of Ketoconazole and an IV (Bolus) Infusion of Eribulin in Patients With Advanced Solid Tumors
Brief Title: Evaluating the Pharmacokinetics and Tolerance of Co-administration of Oral Multiple Dose of Ketoconazole and an IV (Bolus) Infusion of Eribulin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-109
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Cancer
Keywords: Cancer; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — eribulin; Ketoconazole

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Eribulin alone
- Group 2 (Experimental)
  Interventions: Drug: Eribulin plus Ketoconazole

INTERVENTIONS:
Drug: Eribulin alone — Group 1 Cycle 1 (28 days): Eribulin IV 1.4 mg/m^2 alone on Day 1, then eribulin IV 0.7 mg/m^2 plus oral ketoconazole 200 mg on Day 15 and oral ketoconazole 200 mg alone on Day 16. Subsequently, subjects were able to receive eribulin 1.4 mg/m^2 on Days 1 and 8 every 21 days.
  Arms: Group 1
Drug: Eribulin plus Ketoconazole — Group 2 Cycle 1 (28 days): Eribulin IV 0.7 mg/m^2 plus oral ketoconazole 200 mg on Day 1, then oral ketoconazole 200 mg alone on Day 2 and eribulin IV 1.4 mg/m^2 alone on Day 15. Subsequently, subjects were able to receive eribulin 1.4 mg/m^2 on Days 1 and 8 every 21 days.
  Arms: Group 2

SUMMARY:
The purpose of this study is to investigate whether ketoconazole, taken orally, influences the level of eribulin in the blood when the two drugs are given at the same time. The study will enroll patients with solid tumors whose cancer became worse even after standard treatment, or for whom there is no standard treatment available. The study will also investigate whether eribulin given together with ketoconazole is safe (has few side-effects) and is effective against cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically or cytologically confirmed advanced solid tumor that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy).
2. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy ≤ Grade 2 and alopecia.
3. Patients must be aged ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Life expectancy of ≥ 3 months.
6. Patients must have adequate renal function as evidenced by serum creatinine ≤ 2.0 mg/dL (≤ 176 mol/L) or calculated creatinine clearance ≥ 40 mL/minute (min) per the Cockcroft and Gault formula.
7. Patients must have adequate hepatic function as evidenced by bilirubin ≤ 1.5 times the upper limit of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 3 times the ULN, (in the case of liver metastases ≤ 5 times ULN or in the case of bone metastases, the liver specific alkaline phosphatase ≤ 3 times ULN).
8. Patients must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, hemoglobin ≥ 10.0 g/dL or ≥ 6.2 mmol/L (a hemoglobin < 10.0 g/dL or < 6.2 mmol/L is acceptable if it is corrected by growth factor or transfusion), and platelets ≥ 100 x 10^9/L.
9. Patients must be willing and able to comply with the study protocol for the duration of the study.
10. Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have received any of the following treatments within the specified period before eribulin treatment starts:

   1. Chemotherapy, radiation or biological therapy within 2 weeks.
   2. Hormonal therapy within 1 week.
   3. Any investigational drug within 4 weeks.
2. Patients who are receiving anti-coagulant therapy with warfarin or related compounds, other than for line patency and cannot be changed to heparin-based therapy, are not eligible. If a patient is to continue on mini-dose warfarin, then the prothrombin time (PT) or international normalized ratio (INR) must be closely monitored.
3. Patients receiving, at the time the study starts, any medication, dietary supplements or other compounds or substances known to induce or inhibit CYP3A4 activity, with the exception of ketoconazole. A comprehensive list can be found at http://medicine/iupui.edu/flockhart/table.htm.
4. Patients for whom the use of ketoconazole is contraindicated.
5. Patients who are receiving drugs that might influence ketoconazole metabolism.
6. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
7. Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception.
8. Patients whose intestinal absorption is impaired.
9. Severe/uncontrolled intercurrent illness/infection.
10. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association (NYHA) Grade II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia.
11. Patients with organ allografts requiring immunosuppression (not including blood and blood components transfusions).
12. Patients with known positive human immunodeficiency virus (HIV) status.
13. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment with eribulin.
14. Patients with meningeal carcinomatosis.
15. Patients with a hypersensitivity to halichondrin B and/or halichondrin B-like compounds.
16. Patients with pre-existing neuropathy > Grade 2.
17. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jantien Wanders, M.D., Study Director — Eisai Limited
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 center in The Netherlands during the period of Feb 2009 to Jul 2009.
Groups:
- Eribulin Alone First, Then Eribulin Plus Ketoconazole: Eribulin IV 1.4 mg/m^2 alone on Day 1, then eribulin IV 0.7 mg/m^2 plus oral ketoconazole 200 mg on Day 15 and oral ketoconazole 200 mg alone on Day 16 of a 28 day cycle. Subsequently, subjects were able to receive eribulin 1.4 mg/m^2 on Days 1 and 8 every 21 days.
- Eribulin Plus Ketoconazole First, Then Eribulin Alone: Eribulin IV 0.7 mg/m^2 plus oral ketoconazole 200 mg on Day 1, then oral ketoconazole 200 mg alone on Day 2 and eribulin IV 1.4 mg/m^2 alone on Day 15 of a 28 day cycle. Subsequently, subjects were able to receive eribulin 1.4 mg/m^2 on Days 1 and 8 every 21 days.
Period: Cycle 1 Day 1
Arm/Group | Eribulin Alone First, Then Eribulin Plus Ketoconazole | Eribulin Plus Ketoconazole First, Then Eribulin Alone
Started | 6 | 6
Completed | 4 | 6
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Progressive Disease | 1 | 0
Period: Cycle 1 Day 15
Arm/Group | Eribulin Alone First, Then Eribulin Plus Ketoconazole | Eribulin Plus Ketoconazole First, Then Eribulin Alone
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eribulin Alone First, Then Eribulin Plus Ketoconazole | Eribulin Plus Ketoconazole First, Then Eribulin Alone | Total
Number analyzed (Participants) | 6 | 6 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.22) | 62.5 (5.5) | 60.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean (SD) Maximum Observed Concentration (Cmax) of Eribulin
Time Frame: 7 days after dosing on Days 1 and 15
Population: Pharmacokinetic Population: includes all participants in this crossover study who completed PK evaluations and who had Cmax data.
Measure: Mean (Standard Deviation); unit: ng*mL
Groups:
- Eribulin Alone: Eribulin IV 1.4 mg/m^2 alone on Day 1, then eribulin IV 0.7 mg/m^2 plus oral ketoconazole 200 mg on Day 15 and oral ketoconazole 200 mg alone on Day 16 of a 28 day cycle. Subsequently, subjects were able to receive eribulin 1.4 mg/m^2 on Days 1 and 8 every 21 days.
- Eribulin Plus Ketoconazole: Eribulin IV 0.7 mg/m^2 plus oral ketoconazole 200 mg on Day 1, then oral ketoconazole 200 mg alone on Day 2 and eribulin IV 1.4 mg/m^2 alone on Day 15 of a 28 day cycle. Subsequently, subjects were able to receive eribulin 1.4 mg/m^2 on Days 1 and 8 every 21 days.
Arm/Group | Eribulin Alone | Eribulin Plus Ketoconazole
Number analyzed (Participants) | 10 | 10
ng*mL | 207 (73.9) | 106 (33.7)

2. Primary Outcome: Mean (SD) Area Under Concentration Time Curve From Zero to Infinity (AUC 0-oo) of Eribulin
Time Frame: 7 days after dosing on Days 1 and 15
Population: Pharmacokinetic Population: includes all participants in this crossover study who completed PK evaluations and who had AUC (0-oo) data.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Eribulin Alone | Eribulin Plus Ketoconazole
Number analyzed (Participants) | 9 | 7
ng*hr/mL | 971 (371.9) | 482 (241.5)

3. Secondary Outcome: Safety of Eribulin Administered Alone or Coadministered With Oral Ketoconazole, as Measured by Number of Subjects With Adverse Events.
Time Frame: monitored throughout
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Number of participants at risk reflects the Safety Population which included all participants enrolled in this crossover study and received at least a partial dose of study treatment.
Arm/Group | Eribulin Alone | Eribulin Plus Ketoconazole
Serious Adverse Events (participants affected / at risk) | 4/12 | 1/10
Other Adverse Events (participants affected / at risk) | 12/12 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Alone (N=12) | Eribulin Plus Ketoconazole (N=10)
Pyrexia (General disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Metastases to CNS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Alone (N=12) | Eribulin Plus Ketoconazole (N=10)
Nausea (Gastrointestinal disorders) | 9 | 3
Constipation (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 10 | 3
Edema Peripheral (General disorders) | 4 | 1
Pyrexia (General disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinorrhea (Skin and subcutaneous tissue disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1
Weight Decreased (Investigations) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 0
Lacrimation Increased (Eye disorders) | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 0
Herpes Simplex (Infections and infestations) | 2 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No